CLINICAL TRIAL: NCT04547959
Title: Prospective Clinical Study to Evaluate the Efficacy of the Stand-alone Cervical Interbody Cage C-CURVE (Titanium) Manufactured by MEDICREA®
Brief Title: Prospective Clinical Study to Evaluate the Efficacy of the Stand-alone Cervical Interbody Cage C-CURVE ( Titanium) Manufactured by MEDICREA®
Acronym: C-CURVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT220112102
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: C-CURVE , Cervical Interbody Cage; Cervical Disc Disease; Cervical Discopathy
Keywords: cervical disc disease; cervical disc degeneration; C-CURVE , cervical interbody cage

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, non-comparative and interventional post market clinical follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- C-CURVE Titane (Experimental): According the routine practice of the investigator surgeon, the interbody cage C-CURVE in Titane is used
  Interventions: Device: cervical interbody cage C-CURVE

INTERVENTIONS:
Device: cervical interbody cage C-CURVE — ACDF: Anterior Cervical Discectomy and Fusion with a C-CURVE cage

SUMMARY:
This study includes one type of product named C-CURVE which is a Stand-alone Cervical Interbody Cage. This product is available in two materials: PEEK and Titanium.

The C-Curve Cervical Interbody Devices is one single implant used for insertion between two adjacent vertebrae (cervical spine). C-Curve has been designed to restore and/or maintain adequate interbody height, and thus help stabilize one or more cervical levels while fusion occurs. This system has also as objectives to increase of the quality of life, decrease patient's pain and decrease a potential dysphagia (clinical performances). This system must only be used in the cervical spine.

This post-market clinical follow-up (PMCF) study aims to confirm the acceptable benefits/risk profile of the device for the patients and to fill essential requirements to maintain the CE mark through a clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated with C-CURVE TITANIUM (MEDICREA) for one or several levels (3 maximum)
* Cage implanted with the bone graft "OSMOSYS" (MEDICREA) or an auto bone graft from patients
* Patient ≥ 18 years
* Patient affiliated to health care insurance (social security in France)
* Patient who signed an informed consent form
* Patient able and willing to complete a self-administered questionnaire
* Patient able to understand protocol and the planning visit and willing to perform all of them
* Patient with a pathology indicated in the instruction for use of the implant

Exclusion Criteria:

* Patient with no preoperative data available (X-rays, questionnaires)
* Hybrid installation or cervical additional fixation
* Patient contraindicated for X-ray(s) and/or CT-Scan(s)
* Patient with contraindications indicated in the instruction for use of the implant
* Patient judged as non-compliant by the investigator, not unable to come back for the follow-up visits (for example: patient living more than 100 km away).
* Patient who declined to participate to the study or unable to give his consent Vulnerable population as explained in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Fusion of the cervical interbody cage used | 24 months
  Measures the bone fusion thanks to the CTscan

SECONDARY OUTCOMES:
Fusion of the cervical interbody cage used | 6, 12 and 24 months
  Measures the bone fusion thanks to the Xrays
Quality of life with modified SF-12 | Preoperative, and 6, 12 and 24 months postoperative
  Score of the modified SF-12 (to 0 (better) to 100 (worst)
Satisfaction patient | 6, 12 and 24 months
  Score of the PSI (scale: 1/2/3/4 ; 1: Better)
VAS (Pain) | Preoperative, and 6, 12 and 24 months postoperative
  Score of the pain (to 0 (better) to 10 (worst)
NDI(Neck Disability Index) | Preoperative, and 6, 12 and 24 months postoperative
  Score of the pain (to 0 (better) to 50 (worst)
Cervical spinal radiographic parameters (Cobb angle, C2C7 angle, Segmental lordosis/kyphosis, disk height, subsidence, alignment restauration ) for C-CURVE Titanium only | Preoperative, and 6, 12 and 24 months postoperative
  radiographic measurements
Complications | peroperative and 6, 12 and 24 months postoperative
  All Adverse Events related to the study device, instruments and/or the study procedure and all SAEs must be reported
Fusion of the cervical interbody cage used | 6 and 12 months postoperative
  Measures the bone fusion thanks to the CTscan

CONTACTS AND LOCATIONS:
Locations (10):
- CH WAPI, Tournai, Belgium
- France (9):
  - Clinique Belharra, Bayonne
  - Clinique du Parc, Castelnau-le-Lez
  - Groupe Hospitalier La Rochelle-Re-Aunis, La Rochelle
  - Centre de consultations spécialisées de la Sauvegarde, Lyon
  - Centre Orthopédique Santy, Lyon
  - Clinique Clairval, Marseille
  - Clinique de l'Union, Saint-Jean
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - CHRU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alimi M, Njoku I, Hofstetter CP, Tsiouris AJ, Kesavabhotla K, Boockvar J, Navarro-Ramirez R, Hartl R. Anterior Cervical Discectomy and Fusion (ACDF): Comparison Between Zero Profile Implants and Anterior Cervical Plate and Spacer. Cureus. 2016 Apr 17;8(4):e573. doi: 10.7759/cureus.573. PMID 27200226
- [Background] Azab W, Abdel-Razek M, Ali A, Abdelrahman A, Salaheldin W, Nasim K, Attia H, Soliman D. Outcome evaluation of a zero-profile implant for anterior cervical diskectomy with fusion. Turk Neurosurg. 2012;22(5):611-7. doi: 10.5137/1019-5149.JTN.5646-11.2. PMID 23015339
- [Background] Barbagallo GM, Romano D, Certo F, Milone P, Albanese V. Zero-P: a new zero-profile cage-plate device for single and multilevel ACDF. A single institution series with four years maximum follow-up and review of the literature on zero-profile devices. Eur Spine J. 2013 Nov;22 Suppl 6(Suppl 6):S868-78. doi: 10.1007/s00586-013-3005-0. Epub 2013 Sep 24. PMID 24061968
- [Background] Bucci MN, Oh D, Cowan RS, Davis RJ, Jackson RJ, Tyndall DS, Nehls D. The ROI-C zero-profile anchored spacer for anterior cervical discectomy and fusion: biomechanical profile and clinical outcomes. Med Devices (Auckl). 2017 Apr 18;10:61-69. doi: 10.2147/MDER.S127133. eCollection 2017. PMID 28458586
- [Background] Chen Y, Liu Y, Chen H, Cao P, Yuan W. Comparison of Curvature Between the Zero-P Spacer and Traditional Cage and Plate After 3-Level Anterior Cervical Discectomy and Fusion: Mid-term Results. Clin Spine Surg. 2017 Oct;30(8):E1111-E1116. doi: 10.1097/BSD.0000000000000440. PMID 27642818
- [Background] De Leo-Vargas RA, Munoz-Romero I, Mondragon-Soto MG, Martinez-Anda JJ. Locking Stand-Alone Cage Constructs for the Treatment of Cervical Spine Degenerative Disease. Asian Spine J. 2019 Apr 10;13(4):630-637. doi: 10.31616/asj.2018.0234. Print 2019 Aug. PMID 30962412
- [Background] Lee YS, Kim YB, Park SW. Does a zero-profile anchored cage offer additional stabilization as anterior cervical plate? Spine (Phila Pa 1976). 2015 May 15;40(10):E563-70. doi: 10.1097/BRS.0000000000000864. PMID 25955093
- [Background] Li Z, Zhao Y, Tang J, Ren D, Guo J, Wang H, Li L, Hou S. A comparison of a new zero-profile, stand-alone Fidji cervical cage and anterior cervical plate for single and multilevel ACDF: a minimum 2-year follow-up study. Eur Spine J. 2017 Apr;26(4):1129-1139. doi: 10.1007/s00586-016-4739-2. Epub 2016 Aug 23. PMID 27554353
- [Background] Lu Y, Bao W, Wang Z, Zhou F, Zou J, Jiang W, Yang H, Zhang Z, Zhu X. Comparison of the clinical effects of zero-profile anchored spacer (ROI-C) and conventional cage-plate construct for the treatment of noncontiguous bilevel of cervical degenerative disc disease (CDDD): A minimum 2-year follow-up. Medicine (Baltimore). 2018 Feb;97(5):e9808. doi: 10.1097/MD.0000000000009808. PMID 29384883
- [Background] Nambiar M, Phan K, Cunningham JE, Yang Y, Turner PL, Mobbs R. Locking stand-alone cages versus anterior plate constructs in single-level fusion for degenerative cervical disease: a systematic review and meta-analysis. Eur Spine J. 2017 Sep;26(9):2258-2266. doi: 10.1007/s00586-017-5015-9. Epub 2017 Mar 10. PMID 28283840
- [Background] Scholz M, Schelfaut S, Pingel A, Schleicher P, Kandziora F. A cervical "zero-profile" cage with integrated angle-stable fixation: 24-months results. Acta Orthop Belg. 2014 Dec;80(4):558-66. PMID 26280730